CLINICAL TRIAL: NCT05567198
Title: Efficacy of Gonadotropin-releasing Hormone Agonist (GnRHa) in Ovarian Preservation in SLE Subjects Receiving Cyclophosphamide as Determined by Questionnaires
Brief Title: Gonadotropin-releasing Hormone Agonist (GnRHa) in Ovarian Preservation in SLE Subjects Receiving Cyclophosphamide as Determined by Questionnaires
Status: Recruiting | Type: Observational
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001011; 001011-AR
Record Dates: First submitted 2022-10-04; First posted 2022-10-05 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-03-17

CONDITIONS: Systemic Lupus Erythematosus (Sle); Primary Ovarian Insufficiency (Poi)
Keywords: Primary Ovarian Insufficiency (Poi); Nephritis; Neuro-Psychiatric Lupus; Anti-Mullerian Hormone (Amh); Natural History
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Primary Ovarian Insufficiency; Nephritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: SLE patients receiving CYC alone
- Group 2: SLE patients receiving both CYC and leuprolide acetate (GnRH-a)
- Group 3: Control subjects, Age-matched female SLE patients without a history of reproductive disorders

SUMMARY:
Background:

Systemic lupus erythematosus (SLE) is a disease that affects females nine times more often than males. People with SLE are often treated with cyclophosphamide (CYC). But CYC can damage a woman s ovaries; it may cause infertility. A drug called GnRHa is sometimes given to protect the ovaries during CYC therapy. But no one really knows how effective GnRHa treatment is. This natural history survey will compare women who received GnRHa during CYC therapy with those who did not.

Objective:

To find out whether GnRHa can help protect women s ovaries during CYC.

Eligibility:

Women under age 40 years starting CYC treatment with or without GnRHa.

Design:

This study will do 2 things: It will conduct patient surveys. It will collect data from medical records.

Participants will complete a one-time survey. They will answer questions about their menstrual cycle. They will be asked about their history of pregnancy or infertility.

Participants can take the survey in 4 ways:

On paper, sent through the mail.

Online, in a secure web page managed by the NIH.

By phone.

In person, during a routine visit to the NIH clinic.

The survey will take about 30 minutes.

Participants medical records will be reviewed. Researchers will look for data about the participants SLE disease. This may include their symptoms and the results of their blood tests. It may also include the details of prior treatments.

Researchers will also collect data about participants reproductive history. This may include their personal or family history of infertility. It may include any fertility treatments and any sexually transmitted infections.

DETAILED DESCRIPTION:
Study Description: SLE patients with life-threatening lupus manifestations are often treated with cyclophosphamide (CYC), which has known cytotoxic effects on ovarian reserve. Co-administration of Gonadotropinreleasing hormone agonist (GnRHa) is suggested to protect ovaries from the cytotoxic effects of CYC but there is lack of data to support this. We hypothesize that the co-administration of a GnRH agonist for the duration of CYC therapy will exert protective effects on ovarian reserve and function in SLE females. We plan to do a patient survey and a retrospective data collection to compare ovarian function in subjects who received CYC with GnRHa to those who received CYC without GnRHa.

Objectives:

Primary Objective: Determine the effectiveness of GnRH-a in preventing primary ovarian insufficiency (POI) in female SLE patients getting cyclophosphamide treatment.

Secondary Objectives: Determine the effects of SLE disease activity, damage accrual, cumulative dose of cyclophosphamide and other demographic and clinical variables in preventing primary ovarian insufficiency.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:
* INCLUSION CRITERIA: Group 1: SLE patients receiving CYC alone

SLE females <40 years at the beginning of CYC treatment without GnRH-a cotreatment.

-EXCLUSION CRITERIA: Group 1: SLE patients receiving CYC alone

Females >40 years at the beginning of CYC treatment; any females with a prior history of reproductive disorders, infertility, or untreated sexually transmitted infections (STIs).

-INCLUSION CRITERIA: Group 2: SLE patients receiving both CYC and leuprolide acetate (GnRH-a). Leuprolide acetate was injected at a dose of either 3.75 mg/month or 11.25mg/every 3 months.

SLE females <40 years at the beginning of CYC treatment with GnRH-a cotreatment.

-EXCLUSION CRITERIA: Group 2: SLE patients receiving both CYC and leuprolide acetate (GnRH-a). Leuprolide acetate was injected at a dose of either 3.75 mg/month or 11.25mg/every 3 months.

Females >40 years at the beginning of CYC treatment; any females with a prior history of reproductive disorders, infertility, or untreated STIs.

-Group: Control subjects.

Age-matched female SLE patients without a history of reproductive disorders, infertility, or untreated STIs, who have not received CYC either with or without GnRH-a.

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a single-site study which will include women with SLE (diagnosed according to the revised American College of Rheumatology criteria). The participants will be stratified in 3 groups: Group 1: SLE patients receiving CYC alone, Group 2: SLE patients receiving both CYC and leuprolide acetate (GnRH-a), Group 3: Control subjects, Age-matched female SLE patients without a history of reproductive disorders. The subjects screening and retrospective data collection and will be performed by searching electronic medical records for SLE patients treated under SLE Natural History and Pathogenesis Study (Protocol # 94-AR-0066) at the NIH Clinical Center. This protocol and protocol # 94-AR-0066 are under the same PI.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
POI | End of study
  The primary outcome variable is POI, and we want to determine whether GnRH-a coadministration with CYC protects against POI incidence in pre-menopausal SLE females. The age of menopause onset will be collected from previous medical records or survey responses and compared across all three groups. Onset of menopause prior to the age of 40 will be considered POI, whereas menopause onset beyond the age of 40 will be considered natural menopause.

SECONDARY OUTCOMES:
Record Effects of CYC administration with GnRH-a on menstrual cycle | End of study
  - Menses cycles will be classified as either regular (consistently having a period of normal duration each month) or irregular (frequent, infrequent, or absent periods). Classifications of irregular cycle subcategories will be provided, which include polymenorrhea (frequent periods with a cycle length <21 days), oligomenorrhea (infrequent menses with cycle length between 37 to 90 days), or amenorrhea (absence of a period for >90 days). - Menopausal signs and symptoms will include vaginal dryness, hot flashes, chills, sleeping disturbances, night sweats, mood changes, weight gain, loss of breast fullness, thinning hair, or dry skin. - Inability to conceive will be defined as 12 months of trying to conceive without success.
SLE disease activity as measured by SELENA-SLEDAI score at the start of CYC treatment | End of study
  These include SLE disease activity as measured by SELENA-SLEDAI score at the start of CYC treatment, damage index score as measured by SLICC/ACR DI, cumulative CYC dose, and age at the time of beginning CYC.

CONTACTS AND LOCATIONS:
Overall Officials: Sarfaraz A Hasni, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friedman RC, Clarkin JF, Corn R, Aronoff MS, Hurt SW, Murphy MC. DSM-III and affective pathology in hospitalized adolescents. J Nerv Ment Dis. 1982 Sep;170(9):511-21. doi: 10.1097/00005053-198209000-00001. No abstract available. PMID 7108499
- [Background] Kiriakidou M, Cotton D, Taichman D, Williams S. Systemic lupus erythematosus. Ann Intern Med. 2013 Oct 1;159(7):ITC4-1. doi: 10.7326/0003-4819-159-7-201310010-01004. No abstract available. PMID 24081299
- [Background] Stamenovic B. [Effect of increased chloride on the spontaneous release of acetylcholine in the neuromuscular synapses of amphibia poisoned with Clostridium toxin Type A]. Vojnosanit Pregl. 1972 Mar;29(3):139-44. No abstract available. Serbian. PMID 4555317